CLINICAL TRIAL: NCT05296031
Title: Randomized Trial Comparing Drug Eluting Stent Zilver PTX vs Bare Metal Stent Zilver Flex in Critical Limb Ischemia and Treatment of Lesions in Femoral and Popliteal Arteries"
Brief Title: Drug Eluting Stent Zilver PTX vs Bare Metal Stent Zilver Flex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Torbjorn Fransson, Principal Investigator, Consultant Vascular Surgeon, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TF2
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing drug eluting stent Zilver PTX vs Bare metal stent Zilver Flex in critical limb ischemia and treatment of lesions in femoral and popliteal arteries
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Eluting Stent (DES) (Active Comparator): Drug Eluting Stent (DES). Zilver PTX.
  Interventions: Device: Treatment with Zilver PTX Drug Eluting Stent (DES) in femoropopliteal lesions
- Bare Metal Stent (BMS) (Placebo Comparator): Bare Metal Stent (BMS). Zilver Flex
  Interventions: Device: Treatment with Zilver Flex Bare Metal Stent (BMS) in femoropopliteal lesions

INTERVENTIONS:
Device: Treatment with Zilver PTX Drug Eluting Stent (DES) in femoropopliteal lesions — Randomized trial comparing drug eluting stent Zilver PTX vs Bare metal stent Zilver Flex in critical limb ischemia and treatment of lesions in femoral and popliteal arteries
  Arms: Drug Eluting Stent (DES)
Device: Treatment with Zilver Flex Bare Metal Stent (BMS) in femoropopliteal lesions — Randomized trial comparing drug eluting stent Zilver PTX vs Bare metal stent Zilver Flex in critical limb ischemia and treatment of lesions in femoral and popliteal arteries
  Arms: Bare Metal Stent (BMS)

SUMMARY:
Randomized study comparing the results between drug-eluting stents and standard bare metal stents, when treating femoropopliteal lesions in patients with critical limb ischemia.

ELIGIBILITY:
Inclusion Criteria:

Critical limb ischemia RC 4-6

Lesions in superficial femoral artery and popliteal artery (p1 -p2)

Target vessel 4-8mm

At least I 1 vessel runoff to the foot

Age >18 years

Exclusion Criteria:

Pregnancy

Patient disapproval

Age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Freedom from TLR (Target Lesion Revascularization) | 6 months
  Fraction of study subjects without need for retreatment at treatment location
Freedom from TLR (Target Lesion Revascularization) | 12 months
  Fraction of study subjects without need for retreatment at treatment location
Freedom from TLR (Target Lesion Revascularization) | 24 months
  Fraction of study subjects without need for retreatment at treatment location
Open (functioning and not stenosed) vascular reconstruction (Primary Patency) | 12months
  Functioning revascularization without adjunctive measures
Open (functioning and not stenosed) vascular reconstruction (Primary Patency) | 24 months
  Functioning revascularization without adjunctive measures
Event Free Survival | 24 months
  Alive without vascular events